CLINICAL TRIAL: NCT06341621
Title: A Prospective, Randomized, Open-label, Multicenter Phase III Study to Explore Chemotherapy Omission in ER+/HER2-endocrine-sensitive Breast Cancer With 1-3 Positive Lymph Nodes Receiving Extended Adjuvant Abemaciclib
Brief Title: Chemotherapy Omission in ER+/HER2- Breast Cancer With 1-3 Positive Lymph Nodes Receiving Extended Adjuvant Abemaciclib
Acronym: Rainbow
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N071
Record Dates: First submitted 2024-03-16; First posted 2024-04-02 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: adjuvant chemotherapy omission; adjuvant abemeciclib
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Arm 1# endocrine drug plus 3-year abemaciclib without chemotherapy Arm 2# treatment of physician's choice
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endocrine drug plus 3-year abemaciclib without chemo (Experimental): aromatase inhibitors with or without GnRHa plus 3-year lower dose (100mg bid) abemaciclib without chemotherapy.
  Interventions: Drug: 3-year abemaciclib without chemo
- treatment of physician's choice (Active Comparator): treatment of physician's choice, including whether to receive chemotherapy, the chemotherapy regimen and the endocrine therapy regimen.
  Interventions: Drug: treatment of physician's choice

INTERVENTIONS:
Drug: 3-year abemaciclib without chemo — aromatase inhibitors (± ovarian suppression) plus 3-year abemaciclib (100mg bid) without chemotherapy.
  Arms: endocrine drug plus 3-year abemaciclib without chemo
Drug: treatment of physician's choice — treatment of physician's choice including whether to receive chemotherapy, chemotherapy regimen and endocrine therapy regimen.
  Arms: treatment of physician's choice

SUMMARY:
This is a prospective, randomized, open-label, multicenter phase III study to explore chemotherapy omission in ER+/HER2-endocrine-sensitive breast cancer with 1-3 positive lymph nodes receiving extended (3 year) adjuvant abemaciclib

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, multicenter phase III study to explore chemotherapy omission in estrogen receptor (ER)-positive, human epidermal growth factor receptor 2 (HER2)-negative endocrine-sensitive breast cancer with 1-3 positive lymph nodes receiving extended (3 year) adjuvant abemaciclib. In this study, patient eligible will be randomized into either endocrine drug plus 3-year adjuvant abemaciclib without chemotherapy or treatment of physician's choice (TPC).The safety and efficacy of each group will be assessed through invasive disease free survival (iDFS), disease-free survival (DFS), distant disease free survival (DDFS), overall survival (OS) and adverse effects (AE) as graded by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-80 years old;
* Patient has localized invasive breast carcinoma with1-3 positive lymph nodes, T1-T2，and is ER+/HER2- confirmed by histopathology after early breast cancer surgery#HER2-negative breast cancer (based on most recently analyzed biopsy) defined as a negative in situ hybridization test or an Immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (Fluorescence in situ hybridization (FISH), Chromogenic in situ hybridization (CISH) .
* ER≥50%
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 109 /L; platelet count ≥ 100 * 109 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST) ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤

  1×ULN#and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula).
* Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

* Has received neoadjuvant therapy (include chemotherapy, targeted therapy, radiotherapy or endocrine therapy#;
* Has bilateral breast cancer;
* Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
* Has metastatic (Stage 4) breast cancer;
* Has any ≥T3 lesion
* Is pregnant, is breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
* Patients participating in other clinical trials at the same time;
* Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
* Has severe or uncontrolled infection;
* the researchers judged patients to be unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2027-02-25 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Invasive disease free survival | 5 year

SECONDARY OUTCOMES:
disease free survival | 5 year
distant disease free survival | 5 year
overall survival | 5 year
Time Frame: 5 years] 5. adverse effects adverse effects | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhimin Shao, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhimin Cancer Shao, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided